CLINICAL TRIAL: NCT06620172
Title: CT-guided vs Fluoroscopy-guided Trigeminal Ganglion Radiofrequency Thermocoagulation for Idiopathic Trigeminal Neuralgia: A Randomized Controlled Trial
Brief Title: CT-guided vs Fluoroscopy-guided Trigeminal Ganglion Radiofrequency Thermocoagulation for Idiopathic Trigeminal Neuralgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ahmed Awad Bessar, Assistant Professor of Diagnostic and Interventional Radiology, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TN_RFT
Record Dates: First submitted 2024-09-01; First posted 2024-10-01 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Trigeminal Neuralgia; Trigeminal Neuralgia, Idiopathic
Keywords: CT-guided Radiofrequency Thermocoagulation; Fluoroscopy-guided Radiofrequency Thermocoagulation; Idiopathic Trigeminal Neuralgia; Pain Management; Interventional Pain Treatment
MeSH Terms: conditions — Trigeminal Neuralgia; Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Given the specific nature of the interventions, it may not be possible to blind participants or operators; however, to minimize potential bias, outcome assessors will be blinded to the treatment assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT-guided RFT (Experimental): Participants will undergo CT-guided trigeminal ganglion radiofrequency thermocoagulation (RFT) with real-time CT imaging for needle placement and monitoring.
  Interventions: Procedure: CT-guided Radiofrequency Thermocoagulation (RFT)
- Fluoroscopy-guided RFT (Active Comparator): Participants will undergo fluoroscopy-guided trigeminal ganglion radiofrequency thermocoagulation (RFT) with fluoroscopic imaging for needle placement and monitoring.
  Interventions: Procedure: Fluoroscopy-guided Radiofrequency Thermocoagulation (RFT)

INTERVENTIONS:
Procedure: CT-guided Radiofrequency Thermocoagulation (RFT) — Participants in this group will undergo CT-guided trigeminal ganglion radiofrequency thermocoagulation (RFT). The procedure involves real-time CT imaging to guide the placement of the needle and monitor the process.
  Arms: CT-guided RFT
Procedure: Fluoroscopy-guided Radiofrequency Thermocoagulation (RFT) — Participants in this group will undergo fluoroscopy-guided trigeminal ganglion radiofrequency thermocoagulation (RFT). The procedure utilizes fluoroscopic imaging for needle placement and monitoring.
  Arms: Fluoroscopy-guided RFT

SUMMARY:
The goal of this clinical trial is to compare the effectiveness and safety of CT-guided versus fluoroscopy-guided trigeminal ganglion radiofrequency thermocoagulation (TG-RFT) in treating idiopathic trigeminal neuralgia (TN) in adults aged 18 and older.

The main questions it aims to answer are:

* Does CT-guided TG-RFT provide better pain relief compared to fluoroscopy-guided TG-RFT?
* What are the differences in medication consumption between the two methods?
* What are the procedure-related adverse events for both methods?

Investigators will compare CT-guided TG-RFT to fluoroscopy-guided TG-RFT to see if one method is superior in treating idiopathic TN.

Participants will:

* Undergo either CT-guided or fluoroscopy-guided TG-RFT procedure
* Be monitored post-procedure and followed up at 1, 3, and 6 months for pain relief, medication consumption, and adverse events.

DETAILED DESCRIPTION:
This randomized controlled trial aims to compare the efficacy and safety of CT-guided versus fluoroscopy-guided trigeminal ganglion radiofrequency thermocoagulation (TG-RFT) in patients with idiopathic trigeminal neuralgia (TN). Idiopathic TN is characterized by severe, recurrent facial pain, and radiofrequency thermocoagulation is a common interventional treatment option.

Participants eligible for this study will be adults over 18 years old, diagnosed with idiopathic TN based on the International Headache Society criteria, experiencing pain for at least six months with a numeric rating scale (NRS) score greater than 6 despite medical treatment.

Exclusion criteria include vascular compression of the trigeminal nerve by MRI, secondary causes such as multiple sclerosis, trigeminal autonomic cephalalgias, dental or temporomandibular joint pathologies, previous interventional procedures or surgery for TN, coagulopathy, use of antiaggregants and anticoagulants, cardiac pacemaker, renal-hepatic insufficiency, psychiatric illness, malignancy, or infection at the injection site or systemic infection.

Participants will be randomly assigned to either the CT-guided or fluoroscopy-guided RFT group using a computer-generated randomization list. Both procedures will be performed under aseptic conditions with appropriate monitoring and anesthesia. The CT-guided RFT will use real-time CT imaging for needle placement and monitoring, while the fluoroscopy-guided RFT will use fluoroscopic imaging.

The primary outcome measure is pain relief, assessed at 1-, 3-, and 6-months post-procedure using the Numeric Rating Scale (NRS) and Visual Analog Scale (VAS). Secondary outcomes include changes in medication consumption assessed by the Medication Quantification Scale III (MQS III) and the recording of procedure-related adverse events.

This study aims to provide valuable insights into the comparative effectiveness and safety of CT-guided versus fluoroscopy-guided TG-RFT in managing idiopathic TN, potentially guiding future clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Idiopathic trigeminal neuralgia (TN) based on the International Headache Society criteria
* Pain for at least six months and a NRS score greater than 6 despite medical treatment
* Able to provide informed consent.
* Agree to follow the study procedures and attend follow-up visits.

Exclusion Criteria:

* Vascular compression of the trigeminal nerve by MRI and MRI angiography and the presence of secondary causes such as multiple sclerosis
* Trigeminal autonomic cephalalgias accompanied by autonomic symptoms
* Dental or temporomandibular joint pathologies
* Previous interventional procedures or surgery for TN
* Coagulopathy or use of antiaggregants and anticoagulants
* Cardiac pacemaker
* Renal-hepatic insufficiency
* Diagnosis of psychiatric illness
* Malignancy
* Injection site or systemic infection
* Current participation in another clinical trial that could interfere with the outcomes of this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Pain Relief - Numeric Rating Scale (NRS) | Baseline, immediately post-procedure, 1 month, 3 months, and 6 months post-procedure.
  The primary outcome measure will be the level of pain relief, as assessed by the Numeric Rating Scale (NRS), a 0-10 scale where 0 represents "no pain" and 10 represents "worst possible pain.". Pain levels will be recorded at baseline (pre-procedure), immediately post-procedure, and at 1-, 3-, and 6-months post-procedure.
Pain Relief - Visual Analog Scale (VAS) | Baseline, immediately post-procedure, 1 month, 3 months, and 6 months post-procedure.
  Additionally, pain relief will be assessed by the Visual Analog Scale (VAS), a continuous scale ranging from 0 to 100 mm, where 0 represents "no pain" and 100 represents "worst possible pain." Pain levels will be recorded at the same time points: baseline, immediately post-procedure, and at 1-, 3-, and 6-months post-procedure.

SECONDARY OUTCOMES:
Medication Consumption | 6 months post-procedure
  Changes in medication consumption will be assessed using the Medication Quantification Scale III (MQS III) at 6 months post-procedure. This measure will evaluate the impact of the interventions on the need for medications to manage trigeminal neuralgia.
Procedure-related Adverse Events | Immediately post-procedure, 1 month, 3 months, and 6 months post-procedure
  Adverse events related to the interventions will be systematically recorded to evaluate the safety profile of CT-guided versus fluoroscopy-guided trigeminal ganglion radiofrequency thermocoagulation (TG-RFT). Adverse events will be monitored and recorded immediately post-procedure and during follow-up visits at 1, 3, and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Bessar, MD, PhD, Principal Investigator — Assistant Professor of Diagnostic and Interventional Radiology, Zagazig Uni.
Locations (1):
- Zagazig University, Faculty of Medicine, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No
At this time, there is no plan to share individual participant data (IPD) with other researchers. This decision is based on considerations related to patient confidentiality, data privacy concerns, and the absence of a current infrastructure for secure data sharing. The primary results of the study will be published in peer-reviewed journals and presented at scientific conferences, ensuring that the findings are accessible to the broader research community.